CLINICAL TRIAL: NCT00282763
Title: Proprietary Information - Exploratory (Non-confirmatory) Trial
Brief Title: A Research Study to Evaluate the Safety and Effectiveness of MK0686 for the Treatment of Postherpetic Neuralgia (Also Known as PHN or Post Shingles Pain) (0686-005)
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 0686-005; 2005_090
Record Dates: First submitted 2006-01-24; First posted 2006-01-27 (Estimated); Last update posted 2015-11-23 (Estimated); Status verified 2015-11

CONDITIONS: Neuralgia, Postherpetic
MeSH Terms: conditions — Neuralgia, Postherpetic | interventions — methyl 3-chloro-3'-fluoro-4'-(1-(((1-((trifluoroacetyl)amino)cyclopropyl)carbonyl)amino)ethyl)-1,1'-biphenyl-2-carboxylate

INTERVENTIONS:
Drug: MK0686

SUMMARY:
The purpose of this Study is to test the Safety and Effectiveness of MK0686 in relieving neuropathic (chronic) pain as experienced by patients with Postherpetic Neuralgia (Also Know as PHN or Post Shingles Pain).

This is an early phase trial and some specific protocol information is proprietary and not publicly available at this time. (Full information is available to trial participants).

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of postherpetic neuralgia with pain having lasted at least 6 months
* Able to complete study questionnaires, patient diary, and comply with daily study medication
* Patient is not satisfied with current treatment for pain control

Exclusion Criteria:

* Pregnant or nursing female
* History of evidence of a condition that in the opinion of the investigator, may interfere with the study results (e.g., diabetic neuropathy of fibromyalgia) or pose undue risk to undergo the course of medication required by the study (e.g., unstable heart disease, morbid obesity, kidney or liver disease)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2005-12; Primary Completion 2006-08 (Actual); Study Completion 2006-08 (Actual)

PRIMARY OUTCOMES:
proprietary information - exploratory (non-confirmatory) trial

SECONDARY OUTCOMES:
proprietary information - exploratory (non-confirmatory) trial

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC